CLINICAL TRIAL: NCT03582943
Title: Effects of Remote Limb Ischemic Conditioning on Motor Learning in Middle-aged and Older Adults
Brief Title: Effects of RLIC on Motor Learning in Middle-aged and Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Catherine E. Lang, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIHR01HD085930-Aim3; R01HD085930 (NIH)
Record Dates: First submitted 2018-06-18; First posted 2018-07-11 (Actual); Results first posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Adults; Older Adults
Keywords: remote ischemic conditioning, motor learning

STUDY DESIGN:
Intervention Model Description: Single blinded, randomized, controlled trial
Who Masked: Participant
Masking Description: Participants are masked to their group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote limb ischemic conditioning (RLIC) (Experimental): RLIC is achieved via blood pressure cuff inflation to 20 mmHg above systolic blood pressure on the dominant arm. RLIC requires 45 minutes and involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation. RLIC is performed on visits 1-7.
  Interventions: Behavioral: RLIC; Behavioral: Balance training
- Sham conditioning (Sham Comparator): Sham conditioning is achieved via blood pressure cuff inflation to 10 mmHg under diastolic blood pressure on the dominant arm. Sham conditioning requires 45 minutes and involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation. Sham conditioning is performed on visits 1-7.
  Interventions: Behavioral: Sham conditioning; Behavioral: Balance training

INTERVENTIONS:
Behavioral: RLIC — See descriptions under arm/group descriptions. RLIC is delivered for 7 visits, occurring on consecutive weekdays.
  Arms: Remote limb ischemic conditioning (RLIC)
Behavioral: Sham conditioning — See descriptions under arm/group descriptions. Sham conditioning is delivered for 7 visits, occurring on consecutive weekdays.
  Arms: Sham conditioning
Behavioral: Balance training — All participants undergo training on a balance board, learning to hold the board level with equal weight on each leg. This is a motor learning task. Participants perform the balance task for 15, 30-second trials per day at visits 3-7.

SUMMARY:
The purpose of this research is to determine if the beneficial effects of remote limb ischemic conditioning on learning seen in young adults are found in middle-aged and older adults.

DETAILED DESCRIPTION:
Ischemic conditioning is an endogenous phenomenon in which exposing a target organ or tissue to one or more brief episodes of ischemia results in protection of that organ against subsequent ischemia. The effects of ischemic conditioning are not confined within an organ but can be can be transferred from one organ to another, a technique called remote ischemic conditioning. A clinically feasible method for this is remote limb ischemic conditioning (RLIC), where episodes of ischemia and perfusion are induced with a blood pressure cuff placed on the arm.

The overall goal of this line of work is to use ischemic conditioning to enhance learning and outcomes in persons with neurologic injuries. Two previous studies have shown that remote limb ischemic conditioning (RLIC) can enhance learning a motor task in healthy young adults. The next step is to determine which individuals would receive maximum benefit from RLIC before applying these findings to clinical rehabilitation populations such as stroke. Numerous factors, such as age, body mass index (BMI), sex, and cardiovascular comorbidities may influence the response. The current study determines if RLIC can enhance learning in middle-aged and older adults with their burden of co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

1. 40-80 years old
2. Had sufficient cognitive skills to provide informed consent and actively participate.

Exclusion Criteria (determined by self-report):

1. History of a neurological condition, balance impairment, or vestibular disorder.
2. History of attentional disorders (ADD/ADHD) that could affect learning.
3. History of sleep apnea which could confound the effects of RLIC.
4. Presence of lower extremity condition, injury, or surgery that would compromise performance on the balance task.
5. Learning disability, sensory, or communication problem that would prevent completion of the study.
6. History of epilepsy, peripheral vascular disease, or blood diathesis which could contraindicate RLIC.
7. Current intensive weight lifting or interval training exercise which could confound the effects of RLIC.
8. Current substance abuse or dependence.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lang, PT, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, all of the individual participant data after de-identification will be submitted to Washington University data repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication of results.
Access Criteria: Data will be available to anyone who wishes to access it through the Washington University data repository.
URL: https://openscholarship.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited by word-of-mouth and through participant registry. Assessed for eligibility, n = 182. Excluded, n = 100 with n = 33 not meeting criteria, n = 64 declined to participate, and n = 3 pilot participants who were not randomized.
Period: Allocated to Groups
Arm/Group | Remote Limb Ischemic Conditioning (RLIC) | Sham Conditioning
Started | 42 | 40
Completed | 41 | 39
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Intervention and Follow up
Arm/Group | Remote Limb Ischemic Conditioning (RLIC) | Sham Conditioning
Started | 41 | 39
Completed | 37 | 37
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2
Period: Analyzed
Arm/Group | Remote Limb Ischemic Conditioning (RLIC) | Sham Conditioning
Started | 37 | 37
Completed | 33 | 36
Not Completed | 4 | 1
Not completed — Protocol Violation | 4 | 1

BASELINE CHARACTERISTICS:
Population: Only persons who made it through the study (e.g. did not withdraw) and did not have protocol violations were included in the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Remote Limb Ischemic Conditioning (RLIC) | Sham Conditioning | Total
Number analyzed (Participants) | 33 | 36 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (10.5) | 61.8 (9.0) | 61.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 47
  Male | 11 | 11 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 25 | 26 | 51
  Race: African-American | 8 | 10 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 36 | 69
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (4.4) | 26.8 (5.1) | 26.6 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Balance Score
Description: Balance score at the end of training - balance score at baseline, where balance score is the average amount of time in seconds that a participant maintains the stability platform within ±3° of horizontal position during 5 trials of 30 seconds each. Five trials are averaged to form the balance score at each time point.
Time Frame: 1 week
Population: Only participants who completed the entire protocol and did not have a protocol deviation were analyzed.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Remote Limb Ischemic Conditioning (RLIC) | Sham Conditioning
Number analyzed (Participants) | 33 | 36
seconds | 5.55 (4.85) | 4.81 (3.47)
Statistical Analysis 1: Comparison: Remote Limb Ischemic Conditioning (RLIC) vs Sham Conditioning; Test type: Superiority — A priori power analyses was designed to detect at least a 3 second difference in change in balance scores between groups; p = 0.984, Mixed Models Analysis — Test of differences between groups; Mean Difference (Net) = 0.74
Statistical Analysis 2: Comparison: Remote Limb Ischemic Conditioning (RLIC) vs Sham Conditioning; Test type: Superiority; p = .455, Mixed Models Analysis — Test of interaction between age and RLIC vs. sham; Mean Difference (Net) = -0.023
Statistical Analysis 3: Comparison: Remote Limb Ischemic Conditioning (RLIC) vs Sham Conditioning; Test type: Superiority; p = 0.803, Mixed Models Analysis — Test of interaction between sex and RLIC vs. sham conditioning; Mean Difference (Final Values) = 0
Statistical Analysis 4: Comparison: Remote Limb Ischemic Conditioning (RLIC) vs Sham Conditioning; Test type: Superiority; p = 0.233, Mixed Models Analysis — Test of interaction between BMI and RLIC vs. sham conditioning; Mean Difference (Net) = 0.25
Statistical Analysis 5: Comparison: Remote Limb Ischemic Conditioning (RLIC) vs Sham Conditioning; Test type: Superiority — Test of interaction between presence of co-morbidities and RLIC vs. sham conditioning; p = 0.29, Mixed Models Analysis; Mean Difference (Net) = 4.12

ADVERSE EVENTS:
Time Frame: From enrollment through follow-up for a total of 6 weeks
Arm/Group | Remote Limb Ischemic Conditioning (RLIC) | Sham Conditioning
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/36
Other Adverse Events (participants affected / at risk) | 0/33 | 0/36

LIMITATIONS AND CAVEATS:
This was a Phase I study in a small sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT03582943/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT03582943/Prot_SAP_001.pdf